CLINICAL TRIAL: NCT06591754
Title: A Pilotstudy Investigating Feasability, Acceptability and Preliminary Effects of ISTDP (Intensive Short Term Dynamic Psychotherapy) for Patients with Personality Disorder in a Psychiatric Clinic Specialized on Depression, Anxiety and PTSD
Brief Title: Feasibility, Acceptability, and Preliminary Effects of ISTDP for Personality Disorders in a Specialized Psychiatric Clinic
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Stockholm University (Other)
Responsible Party: Principal Investigator, Maria Bragesjo, PhD and licensed psychologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04361-01
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Personality Disorder
Keywords: Personality disorder; ISTDP; Intensive Short-Term Dynamic Psychotherapy
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ISTDP (Experimental): ISTDP combined group- and individual therapy
  Interventions: Behavioral: ISTDP

INTERVENTIONS:
Behavioral: ISTDP — Both the individual therapy and the group therapy is based on ISTDP (Intensive Short-Term Dynamic Psychotherapy), an affect-focused psychodynamic therapy method. The therapy focus on the relationship between feelings, anxiety and dysfunctional emotion regulation (i.e. defenses). The purpose is to increase the capacity of anxiety regulation in the patient and to help the patient identify the dysfunctional patterns developed to avoid internal stress and then gradually approach previously warded of feelings. The individual therapy consists of 25 weekly sessions. The group treatment consists of 18 weekly sessions and is structured in three phases. Phase one: Psychoeducation about anxiety and exercises in anxiety regulation. Phase two: patients takes turn to observe their own anxiety and defenses together with a therapist. Phase three: Every session two patients will work with a chosen problem and identify defenses, anxiety and feelings together with a therapist in front of the group.

SUMMARY:
The primary objective of this study is to evaluate the feasibility and acceptability of a 25-week combined group and individual therapy program using Intensive Short-Term Dynamic Psychotherapy (ISTDP) for patients diagnosed with personality disorders. The secondary objective is to investigate preliminary effects of the treatment in terms of reducing symtoms of depression, anxiety and emotion regulation difficulties.

DETAILED DESCRIPTION:
The investigators vill investigate a 25-week treatment with ISTDP that consists of both weekly group- and individual therapy for patients diagnosed with personality disorder in a psychiatric clinic specialized on depression, anxiety and PTSD. The feasibility and acceptability and preliminary effects will be evaluated using a within-group design with repeated measures and qualitative interviews. Patients will be recruited from the clinic and the main inclusion criteria is that the patient have a personality disorder diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Personality disorder diagnosis (Clinical assessment using STIP-5) Speaks Swedish fluently

Exclusion Criteria:

Autism or intellectual disability Borderline, antisocial or narcissistic personality disorder diagnosis Need for interpreter Urgent social misery Psychotic disorder High suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients experience of, and satisfaction with, the treatment assessed through qualitative interviews | Immediately after treatment completion
  Patients experience of, and satisfaction with, the treatment assessed through qualitative interviews
Depression symtoms | Baseline, weekly throughout treatment, immediately after treatment completion and 6-month follow-up
  Depression symtoms will be measured with Patient Health Questionnaire (PHQ-9; (Kroenke et al., 2001)
Participants satisfaction with treatment assessed with the Client Satisfaction Questionnaire (CSQ-8) | Immediately after treatment completion (25 weeks)
  Participants satisfaction with treatment assessed with the Client Satisfaction Questionnaire (CSQ-8)
Adverse events related to the treatment | From start of treatment up to. 6 month follow up.
  Adverse events related to the treatment
Number of individual sessions attended during the treatment | Throughout the treatment period, up to 25 weeks
  Number of individual sessions attended during the treatment
Number of group sessions attended during the treatment | Throughout the treatment period, up to 25 weeks
  Number of group sessions attended during the treatment
Number of dropouts | Throughout the treatment period, up to 25 weeks
  Number of dropouts
Total number of sessions attended during the treatment | Throughout the treatment period, up to 25 weeks
  Total number of sessions attended during the treatment

SECONDARY OUTCOMES:
Fear of negative emotions | Change from baseline to post-treatment (25 weeks) and follow up 6 months after treatment.
  Fear of negative emotion scale (Gilbert et al., 2014) for assessing fear and avoidance of negative feelings.
Anxiety symtoms | Change from baseline to immediately after treatment completion (25 weeks) and follow up 6 months after treatment.
  Generalized Anxiety Disorder-7 (GAD-7; Spitzer et al., 2006) for assessing anxiety symtoms.
Emotions regulation difficulties | Change from baseline to immediately after treatment completion (25 weeks) and follow up 6 months after treatment.
  Difficulties in Emotion Regulation Scale (DERS-16; Bjureberg et al., 2016) for assessing difficulties with emotions regulation.
Severity of personality disorder | Change from baseline to immediately after treatment completion (25 weeks) and follow up 6 months after treatment.
  The Standardized Assessment of Severity of Personality Disorders (SASPD; Olajide et al., 2018) for assessing degree of personality disorder.
Symtoms of Borderline Personality disorder | Change from baseline to immediately after treatment completion (25 weeks) and follow up 6 months after treatment.
  Borderline Symtom List (BLS-23; Bohus et al., 2008) for assessing symtoms of Borderline personality disorder.
Severity of personality disorder | Change from baseline to immediately after treatment completion (25 weeks) and follow up 6 months after treatment.
  Levels of Personality Functioning Brief Form (LPFS-BF; Weekers et al., 2019) for assessing degree of personality disorder.
Quality of life | Change from baseline to immediately after treatment completion (25 weeks) and follow up 6 months after treatment.
  Brunnsviken Brief Quality of life (Lindner et al., 2016) for assessing quality of life.
Quality of life | Change from baseline to immediately after treatment completion (25 weeks) and follow up 6 months after treatment.
  EuroQol-5D (EQ5D; Balestroni, Gianluigi, & Bertolotti, 2015) for assessing quality of life.
Working alliance | Weekly throughout treatment , up to 25 weeks
  Session Alliance Inventory (SAI; Falkenström et al., 2015) for assessing the working alliance with the therapist
Emotional activation during therapy | Weekly throughout treatment, up to 25 weeks
  Emotional Experience Self Report (Fisher et al., 2016) for assessing the degree of emotional activation during the session.

CONTACTS AND LOCATIONS:
Locations (1):
- Affektiva, ångest och traumaprogrammet, Psykiatri Sydväst, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The raw data collected in the study can be made available on a group level given that the request comply with Swedish and EU laws regulating protection of identifiable data.